CLINICAL TRIAL: NCT01700036
Title: A Pilot Study of Alpha-1-Antitrypsin (AAT) in Steroid Refractory Acute Graft vs Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: CSL Behring (Industry); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: umcc 2012.043; HUM 67889 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): Alpha-1-Antitrypsin (AAT) for the treatment of Steroid Refractory Acute Graft vs Host Disease.
  Interventions: Drug: Alpha-1-Antitrypsin (AAT)

INTERVENTIONS:
Drug: Alpha-1-Antitrypsin (AAT) — AAT (Zemaira) will be administered at a dose of 60mg/kg (actual weight) on D1, 4, 8, 12, 16, 20, 24, and 28. A second course of treatment will not be given.
  Other Names: Zemaira

SUMMARY:
This clinical trial will study the safety and efficacy of using the drug Zemaira, an Alpha 1-Antitrypsin (AAT) medication (also known as an Alpha1-Proteinase Inhibitor [Human]) for the treatment of steroid refractory GVHD.

For bone marrow transplant patients, the most common, serious complication is Graft vs Host Disease (GVHD), which at its most severe is a life-threatening, complication and a significant cause of treatment related death, following stem cell transplantation. GVHD is a major obstacle to the overall success of transplant treatment, a strategy that would otherwise provide the possibility of a cure for patients with blood cancers or severe blood disorders. GVHD primarily affects the skin, gut, and liver of the recipient, and involves the interaction of the recipient's (the host's) cells and tissues with the donor's immune system cells that see the host tissues as foreign, and attack the host's cells resulting in tissue and organ damage.

The severity of acute GvHD ranges from mild to severe, and for patients who don't respond to steroid therapy, the complication is nearly always fatal, either from organ damage or opportunistic infection as a consequence of high dose, steroid treatments.

There is currently no known effective therapy for patients with acute graft vs host disease that's refractory (nonresponsive) to steroid therapy. As stated earlier,the overwhelming majority of these patients may ultimately die from infection. The incidence of acute GvHD that requires intervention, is higher for unrelated donor transplants, the most common treatment option available, and therefore, these patients are at higher risk for treatment related complications from GVHD. Approximately 20,000 unrelated donor transplants are performed each year. The magnitude of this problem then is significant for patients who otherwise might be cured of their blood cancer or disease.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients must have clinical evidence* of steroid-refractory acute Graft vs Host Disease (any organ) defined as one of the following:

  * No change or progression in the stage of skin GvHD after at least 1 week of 2mg/kg/day methylprednisolone (or po equivalent)
  * lack of response of visceral (liver, GI) GvHD despite treatment with 2mg/kg/day methylprednisolone for at least 72h.
  * progression of visceral GvHD despite treatment with 2mg/kg/day methylprednisolone for at least 48h
  * visceral GvHD progressing to stage 4 after 24h of 2mg/kg/d methylprednisolone
  * Patients with protracted acute GvHD who have not responded to at least 0.5mg/kg/d of prednisone are considered eligible.
* Ability to understand and the willingness to sign a written informed consent document.
* * As GvHD is a clinical diagnosis, and patients will have already been initiated on steroid therapy at the discretion of the attending physician, tissue confirmation of refractory GvHD by biopsy is not required for entry to this study. It is anticipated that most, but not all, patients will have undergone tissue confirmation of the initial diagnosis of GvHD; however lack of tissue confirmation for this clinical syndrome is not exclusionary.

Exclusion Criteria:

* As patients with steroid refractory acute GvHD are quite ill with multiple abnormal labs and organ dysfunction, there are no explicit laboratory values or degree of organ dysfunction that specifically preclude enrollment on this study. Baseline lab studies will be obtained and followed throughout this trial as the standard of care for patients with GvHD.
* Pregnancy or Nursing Mother
* Vasopressor requirement
* Patients may not be receiving any other investigational agents for the treatment of GvHD at time of study entry or at any time while on study or be on another investigational agent that can impact on the primary clinical outcome analyses or has known pharmacodynamics or pharmacokinetic effects on AAT.
* Patients with known antibodies to IgA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2016-10 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavan Reddy, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan

REFERENCES:
- [Derived] Magenau JM, Goldstein SC, Peltier D, Soiffer RJ, Braun T, Pawarode A, Riwes MM, Kennel M, Antin JH, Cutler CS, Ho VT, Alyea EP 3rd, Parkin BL, Yanik GA, Choi SW, Lewis EC, Dinarello CA, Koreth J, Reddy P. alpha1-Antitrypsin infusion for treatment of steroid-resistant acute graft-versus-host disease. Blood. 2018 Mar 22;131(12):1372-1379. doi: 10.1182/blood-2017-11-815746. Epub 2018 Feb 2. PMID 29437593

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 59 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients That Respond to Treatment
Description: To estimate the proportion of patients with steroid refractory acute Graft vs Host Disease) GvHD who respond (achieve either PR or CR) to Alpha-1 Antitrypsin (AAT) at a dose of 60mg/kg twice weekly for 8 doses
  Partial Response (PR) is defined as a decrease of at least one grade in the severity of GVHD without deterioration of any organ systems by d28 of therapy.
  Complete Response (CR) is defined as the resolution of all manifestations of GVHD by d28 of treatment. All organs must have a Stage 0.
Time Frame: 4 weeks
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Treatment Arm: Alpha-1-Antitrypsin (AAT): AAT (Zemaira) will be administered at a dose of 60mg/kg (actual weight) on D1, 4, 8, 12, 16, 20, 24, and 28.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
percentage of patients | 65 [48 to 79]

2. Secondary Outcome: Percentage of Patients Who Achieve a Complete Response to Treatment
Description: To estimate the proportion of patients in complete remission without additional therapy at four weeks after the last dose of AAT
  Complete remission is defined as the resolution of all manifestations of GVHD by d28 of treatment. All organs must have a Stage 0.
Time Frame: 4 weeks
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
percentage of patients | 35 [21 to 52]

3. Secondary Outcome: Percentage of Patients With Documented Infection
Description: To estimate the incidence of infection during and following treatment of steroid refractory acute GVHD with AAT
Time Frame: 30 days
Measure: Number; unit: percentage of patients
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
percentage of patients | 32.5

4. Secondary Outcome: The Percentage of Patients Alive at 6 Months for Patients in CR or PR
Description: Survival at 6 months in patients receiving AAT treatment for steroid refractory acute GVHD for patients that achieved a CR or PR.
  Partial Response (PR) is defined as a decrease of at least one grade in the severity of GVHD without deterioration of any organ systems by d28 of therapy.
  Complete Response (CR) is defined as the resolution of all manifestations of GVHD by d28 of treatment. All organs must have a Stage 0.
Time Frame: 6 months
Population: 40 patients were enrolled and 26 patients achieved a CR or PR.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment Arm
Number analyzed (Participants) | 26
percentage of patients | 50 [34 to 73]

5. Secondary Outcome: Mean Fold Change in Plasma Biomarkers
Description: The fold change in levels of plasma biomarkers IL-6, TNF-alpha and ST2 will be measured pre-treatment and after the administration of AAT treatment for steroid refractory GvHD.
Time Frame: Baseline, 2 weeks, and 4 weeks
Measure: Mean (Standard Error); unit: fold change from baseline
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
fold change from baseline
  IL-6 Fold Change at 2 weeks | 6.3 (3.6)
  IL-6 Fold Change at 4 weeks | 4 (1.9)
  TNF-alpha Fold Change at 2 weeks | 1.7 (0.8)
  TNF-alpha Fold Change at 4 weeks | 1.1 (0.2)
  ST2 Fold Change at 2 weeks | 1.2 (0.4)
  ST2 Fold Change at 4 weeks | 1.5 (0.7)

6. Secondary Outcome: Mean Plasma Levels for Alpha-1-Antitrypsin (AAT)
Description: Plasma levels of Alpha-1-Antitrypsin(AAT)will be measured.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Treatment Arm
Number analyzed (Participants) | 40
mg/dl
  AAT levels at two weeks | 196.8 (11.91)
  AAT levels at 4 weeks | 214.8 (18.62)

ADVERSE EVENTS:
Time Frame: Patients will be followed for adverse events for 30 days after the last dose of the study drug.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 8/40
Serious Adverse Events (participants affected / at risk) | 11/40
Other Adverse Events (participants affected / at risk) | 31/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=40)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Immune system disorder (Immune system disorders) | 2 (2)
Bladder infection (Infections and infestations) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=40)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3)
Fever (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 1 (1)
Immune system disorder (Immune system disorders) | 2 (2)
Bladder infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 11 (16)
Kidney infection (Infections and infestations) | 1 (2)
Lung infection (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 6 (6)
Lymphocyte count decreased (Investigations) | 5 (6)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 5 (7)
White blood cell decreased (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes